CLINICAL TRIAL: NCT02661854
Title: Double Blind, Placebo-controlled, Dose Finding, Prospective, Multicenter Clinical Trial for the Treatment of Rhinitis/Rhinoconjunctivitis Against a Mixture of Dermatophagoides Pteronyssinus and Dermatophagoides Farinae Allergen Extract
Brief Title: Dose Finding for the Treatment of Rhinitis/Rhinoconjunctivitis Against Mite Allergy
Acronym: MM09
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: MM09-SIT-013; 2015-000820-27 (EudraCT Number)
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Rhinitis; Rhinoconjunctivitis
Keywords: Rhinitis / Rhinoconjunctivitis; Vaccine; Immunotherapy; Mite; Allergy
MeSH Terms: conditions — Rhinitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- MM09 Mannosylated 5.000 subcutaneous (Experimental): 5.000 MTU/ml of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MM09 Mannosylated 5.000 subcutaneous; Biological: Sublingual placebo
- MM09 Mannosylated 10.000 subcutaneous (Experimental): 10.000 MTU/ml of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MM09 Mannosylated 10.000 subcutaneous; Biological: Sublingual placebo
- MM09 Mannosylated 30.000 subcutaneous (Experimental): 30.000 MTU/ml of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MM09 Mannosylated 30.000 subcutaneous; Biological: Sublingual placebo
- MM09 Mannosylated 50.000 subcutaneous (Experimental): 50.000 MTU/ml of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MM09 Mannosylated 50.000 subcutaneous; Biological: Sublingual placebo
- MM09 Mannosylated 5.000 sublingual (Experimental): 5.000 MTU/ml of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MM09 Mannosylated 5.000 sublingual; Biological: Subcutaneous placebo
- MM09 Mannosylated 10.000 sublingual (Experimental): 10.000 MTU/ml of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MM09 Mannosylated 10.000 sublingual; Biological: Subcutaneous placebo
- MM09 Mannosylated 30.000 sublingual (Experimental): 30.000 MTU/ml of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MM09 Mannosylated 30.000 sublingual; Biological: Subcutaneous placebo
- MM09 Mannosylated 50.000 sublingual (Experimental): 50.000 MTU/ml of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MM09 Mannosylated 50.000 sublingual; Biological: Subcutaneous placebo
- Placebo Sublingual Placebo subcutaneous (Placebo Comparator): Sublingual and subcutaneous placebo.
  Interventions: Biological: Subcutaneous placebo; Biological: Sublingual placebo

INTERVENTIONS:
Biological: MM09 Mannosylated 5.000 subcutaneous — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 5.000 MTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Other Names: Manano
  Arms: MM09 Mannosylated 5.000 subcutaneous
Biological: MM09 Mannosylated 10.000 subcutaneous — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 10.000 MTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Arms: MM09 Mannosylated 10.000 subcutaneous
Biological: MM09 Mannosylated 30.000 subcutaneous — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 30.000 MTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Arms: MM09 Mannosylated 30.000 subcutaneous
Biological: MM09 Mannosylated 50.000 subcutaneous — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 50.000 MTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Arms: MM09 Mannosylated 50.000 subcutaneous
Biological: MM09 Mannosylated 5.000 sublingual — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 5.000 MTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MM09 Mannosylated 5.000 sublingual
Biological: MM09 Mannosylated 10.000 sublingual — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 10.000 MTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MM09 Mannosylated 10.000 sublingual
Biological: MM09 Mannosylated 30.000 sublingual — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 30.000 MTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MM09 Mannosylated 30.000 sublingual
Biological: MM09 Mannosylated 50.000 sublingual — Mixture of the following mites: Dermatophagoides pteronyssinus and Dermatophagoides farinae, allergen extract with a concentration of 50.000 MTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MM09 Mannosylated 50.000 sublingual
Biological: Subcutaneous placebo — Comparison between placebo and active group
  Arms: MM09 Mannosylated 10.000 sublingual; MM09 Mannosylated 30.000 sublingual; MM09 Mannosylated 5.000 sublingual; MM09 Mannosylated 50.000 sublingual; Placebo Sublingual Placebo subcutaneous
Biological: Sublingual placebo — Comparison between placebo and active group
  Arms: MM09 Mannosylated 10.000 subcutaneous; MM09 Mannosylated 30.000 subcutaneous; MM09 Mannosylated 5.000 subcutaneous; MM09 Mannosylated 50.000 subcutaneous; Placebo Sublingual Placebo subcutaneous

SUMMARY:
The purpose of the study is to evaluate the more efficient dose for the treatment of rhinitis/rhinoconjunctivitis against mite allergy

DETAILED DESCRIPTION:
Double blind placebo-controlled study. The subjects will receive medication during 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Positive suggestive clinical history of intermittent or persistent moderate to severe rhinitis /rhinoconjunctivitis, with or without moderate asthma, due to Dermatophagoides pteronyssinus and/or Dermatophagoides farinae allergy
* Subjects with a positive skin prick-test (wheal sixe >6 mm diameter)
* Specific immunoglobulin E against house dust mites >10 kU/L and whose determination does not exceed 6 months prior to the inclusion visit
* Age between 12 and 65 years
* Both genders
* Subjects capable of giving informed consent
* Subjects capable of complying with the dosing regimen
* Subjects that have not received immunotherapy in the last 5 years
* Subjects presenting sensitization to another aeroallergens, but that is considered clinically not relevant or no clinical interference with the nasal provocation test.

Exclusion Criteria:

* Subjects outside of the age range.
* Subjects who have previously received immunotherapy for the treatment of the allergic rhinitis/rhinoconjunctivitis due to mites and other allergens in the last 5 years.
* Subjects that immunotherapy may be an absolute contraindication according to the criteria of the immunotherapy Committee of the Spanish society of Allergy and Clinical Immunology, and of the European Allergy and Clinical Immunology Immunotherapy Subcommittee may also include.
* Subjects with important symptoms of rhinoconjunctivitis /bronchial asthma in which the suspension of the systemic antihistamine treatment is contraindicated.
* Subjects with persistent severe or not controlled asthma , with a forced expiratory volume (FEV) < 70 respect to the reference value in spite of the appropriate pharmacological treatment at the time of the inclusion in the trial.
* Subjects that have required oral corticosteroids in the 12 weeks previous to the inclusion in the trial.
* Subjects that have previously submitted a serious secondary reaction during the skin prick test
* Subjects in treatment with beta blockers.
* Unstable subjects from the clinical point of view (respiratory infection, febrile, acute urticaria, etc.) at the time of the inclusion in the clinical trial
* Subject with chronic urticaria in the last 2 years or hereditary angioedema.
* Subjects that have some pathology (hyperthyroidism, hypertension, heart disease, etc.) is contraindicated.
* Subjects with any other disease not associated with the rhinitis/rhinoconjunctivitis, but of potential severity and that could interfere with treatment and follow-up (epilepsy, psychomotor deterioration, diabetes, malformations, multi-operated, kidney diseases,...).
* Subjects with autoimmune disease (lupus, thyroiditis, etc.), tumor or with diagnosis of immunodeficiency diseases.
* Subject whose status prevents him from providing cooperation and or which present severe psychiatric disorders.
* Subject with known allergy to other components of the vaccine different from mites allergen extract.
* Subjects with lower airway diseases other than asthma such as emphysema or bronchiectasis.
* Direct investigator's relatives.
* Pregnant or women at risk of pregnancy and breastfeeding women.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Concentration required to elicit a positive response after nasal provocation test (NPT) | 4 months
  Change in the threshold concentration of mite allergen extract, measured in Histamine Equivalent Prick per ml (HEP/ml), needed to trigger a positive response after nasal provocation test (NPT) assessed by acoustic rhinometry.
  This will be compared between the beginning and end of the trial and among active groups and placebo.

SECONDARY OUTCOMES:
Dose finding skin prick test | 4 months
  Comparison between the beginning and end of the trial and among active groups and placebo
Number of participants with treatment-related adverse events as assessed by MM09-SIT-013 | 4 months
  Comparison between the beginning and end of the trial and among active groups and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mª Dolores Hernández, PhD; MD, Principal Investigator; Pilar Alba, PhD; MD, Principal Investigator; Carmen Pérez, PhD; MD, Principal Investigator; Javier Montoro, PhD; MD, Principal Investigator; Antonio de Mateo, PhD; MD, Principal Investigator; David El-Qutob, PhD; MD, Principal Investigator; Javier Fernández, PhD; MD, Principal Investigator; Vicente Jover, PhD; MD, Principal Investigator; Isabel Flores, PhD; MD, Principal Investigator; Mónica Antón, PhD; MD, Principal Investigator; Carmen Andreu, PhD; MD, Principal Investigator; Luis Angel Navarro, PhD; MD, Principal Investigator; Ángel Ferrer, Principal Investigator; Antonio Nieto, PhD; MD, Study Director
Locations (14):
- Spain (14):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Del Vinalopo, Elche, Alicante
  - Hospital General Universitario de Elda-Virgen de La Salud, Elda, Alicante
  - Hospital Vega Baja Orihuela, Orihuela, Alicante
  - Hospital Universitari de Castelló, Castellon, Castellón
  - Hospital de La Plana, Vila-real, Castellón
  - Hospital de Manises, Manises, Valencia
  - Hospital Lluis Alcanyis de Xátiva, Xátiva, Valencia
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Vithas Internacional Medimar, Alicante
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - HOSPITAL UNIVERSITARI I POLITÈCNIC LA FE Adults, Valencia
  - HOSPITAL UNIVERSITARI I POLITÈCNIC LA FE child, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soria I, Lopez-Relano J, Vinuela M, Tudela JI, Angelina A, Benito-Villalvilla C, Diez-Rivero CM, Cases B, Manzano AI, Fernandez-Caldas E, Casanovas M, Palomares O, Subiza JL. Oral myeloid cells uptake allergoids coupled to mannan driving Th1/Treg responses upon sublingual delivery in mice. Allergy. 2018 Apr;73(4):875-884. doi: 10.1111/all.13396. Epub 2018 Jan 31. PMID 29319882
- [Background] Manzano AI, Javier Canada F, Cases B, Sirvent S, Soria I, Palomares O, Fernandez-Caldas E, Casanovas M, Jimenez-Barbero J, Subiza JL. Structural studies of novel glycoconjugates from polymerized allergens (allergoids) and mannans as allergy vaccines. Glycoconj J. 2016 Feb;33(1):93-101. doi: 10.1007/s10719-015-9640-4. Epub 2015 Nov 25. PMID 26603537
- [Background] Sirvent S, Soria I, Cirauqui C, Cases B, Manzano AI, Diez-Rivero CM, Reche PA, Lopez-Relano J, Martinez-Naves E, Canada FJ, Jimenez-Barbero J, Subiza J, Casanovas M, Fernandez-Caldas E, Subiza JL, Palomares O. Novel vaccines targeting dendritic cells by coupling allergoids to nonoxidized mannan enhance allergen uptake and induce functional regulatory T cells through programmed death ligand 1. J Allergy Clin Immunol. 2016 Aug;138(2):558-567.e11. doi: 10.1016/j.jaci.2016.02.029. Epub 2016 Apr 13. PMID 27177779
- [Background] Soria I, Alvarez J, Manzano AI, Lopez-Relano J, Cases B, Mas-Fontao A, Canada FJ, Fernandez-Caldas E, Casanovas M, Jimenez-Barbero J, Palomares O, Vinals-Florez LM, Subiza JL. Mite allergoids coupled to nonoxidized mannan from Saccharomyces cerevisae efficiently target canine dendritic cells for novel allergy immunotherapy in veterinary medicine. Vet Immunol Immunopathol. 2017 Aug;190:65-72. doi: 10.1016/j.vetimm.2017.07.004. Epub 2017 Jul 23. PMID 28778325